CLINICAL TRIAL: NCT03175783
Title: Use of Wearable Activity Tracker to Monitor and Increase Mobility for Elderly Undergoing Abdominal Surgery: A Randomized Control Trial
Brief Title: Use of Wearable Activity Tracker in Elderly Undergoing Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Wong Koh Ging, Doctor, University of Malaya
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 36100
Record Dates: First submitted 2017-05-27; First posted 2017-06-05 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Fitness Trackers; Early Ambulation; Surgery; Health Services for the Aged

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Treatment group will receive intervention by putting on Fitbit Zip activity tracker with automatic step counts feedback throughout the study.
  Interventions: Device: Fitbit Zip Activity Tracker
- Control Group (Sham Comparator): Control group will be put on intervention with same Fitbit Zip activity tracker but without automatic feedback for same duration of intervention.
  Interventions: Device: Fitbit Zip Activity Tracker

INTERVENTIONS:
Device: Fitbit Zip Activity Tracker — Subjects from both treatment and control group will be put on wristband starting from one week before the scheduled operation until 7 post-operative days. Patients will be instructed to wear the wristband continuously 24 hours per day except during water based activity. The treatment group will receive normal wristband with indicator showing steps count, distance, and calories. Meanwhile, the control group will receive Fitbit Zip with a display covered with adhesive tape and will not receive automatic feedback on the mobility from the device.

SUMMARY:
Early mobilization is an important element in Enhanced Recovery After Surgery (ERAS). It reduces risk of conditions which are related to prolonged bed rest such as deep vein thrombosis, lung atelectasis, pneumonia, and sacral sore. (Appelboom, Taylor et al. 2015) It is also associated with shortened length of hospital stay, improved survival, and reduction in health care cost.

However, "early mobilization" was not defined consistently in previous study. Some authors recommend patients to get out of bed and ambulate on the day of operation while others define as getting out of bed more than 2 hours on day of operation and up to 8 hours on second post-operative day. (Wolk, Meissner et al. 2017) The inconsistency in definition is partly due to the inability to quantify patients' mobility which is usually self-reported by patients and is subjective.(Eva van der Meij 2017) This is especially true for elderly patient in whom preoperative mobility varies significantly between individuals. For this reason, the approach of early mobilization in elderly should be goal directed and individualized according to their preoperative mobility and functional status.

The aim of current study is to monitor and motivate elderly patients undergoing abdominal surgery to increase postoperative mobilization by using Fitbit Zip activity tracker.

DETAILED DESCRIPTION:
This is a randomized, controlled, single center trial comparing the use of activity tracker with and without automatic feedback in improving postoperative mobility of elderly patients undergoing abdominal surgery.

Selected subjects will be randomized into treatment and control groups in a ratio of 1:1.

Patients will be randomized upon enrollment using computer generated random assignment. Treatment group will be put on activity tracker device (Fitbit Zip) with automatic step counts feedback throughout the study. Meanwhile, control group will be put on same activity tracker without automatic feedback for same duration of intervention. The Fitbit Zip tracker (Fitbit Inc, San Francisco, California USA) is a validated commercially available activity tracker and its use has been proven accurate in elderly patients.

Subjects from both treatment and control group will be put on wristband starting from one week before the scheduled operation until 7 post-operative days. Patients will be instructed to wear the wristband continuously 24 hours per day except during water based activity. The treatment group will receive normal wristband with indicator showing steps count, distance, and calories. Meanwhile, the control group will receive Fitbit Zip with a display covered with adhesive tape and will not receive automatic feedback on the mobility from the device.

At the end of the intervention, all the data will be retrieved from the Fitbit Zip via Fitbit Connect software 2.0. On top of that, data on patients' demographic, types of operation, operative findings, length of hospital stay and postoperative complication will also be recorded in case report form.

ELIGIBILITY:
Inclusion Criteria:

* Adult age >60 years old
* Patients electively scheduled for abdominal surgery includes upper gastro-intestinal surgery (subtotal gastrectomy, partial gastrectomy), colorectal surgery (hemicolectomy, anterior resection, sigmoidectomy, abdominal perineal resection), and hepatobiliary surgery ( pancreatectomy, cholecystectomy, hepatectomy)
* Able to provide informed consent

Exclusion Criteria:

* Cognitive impairment
* Neurological deficit which requires assistance in mobilization (e.g stroke, post limb amputation)
* Emergency surgery
* Prolonged ventilation >24 hours
* Prolonged stay in ICU >48 hours
* Lack of compliance to wearing wrist band
* Allergic to wristband

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative mobility measured by mean step counts | 14 days
  Comparing mean step counts between treatment and control group

SECONDARY OUTCOMES:
Percent change in postoperative mobility | 14 days
  Percentage of step counts achieved by subject post-operatively is compared with subject's baseline step counts
Effect of activity tracker with automatic feedback on length of hospital stay | up to one month
  Compare the length of hospital stay between the treatment group and control group
Number of patients with post operative complications | up to one month
  Rate of complications related to immobilisation (deep vein thrombosis, atelectasis, pneumonia, decubitus ulcer, pulmonary embolism, bedsore) are compared between treatment and control group

CONTACTS AND LOCATIONS:
Overall Officials: Wong Koh Ging, MD, Principal Investigator — University of Malaya
Locations (1):
- Sarawak General Hospital, Kuching, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appelboom G, Taylor BE, Bruce E, Bassile CC, Malakidis C, Yang A, Youngerman B, D'Amico R, Bruce S, Bruyere O, Reginster JY, Dumont EP, Connolly ES Jr. Mobile Phone-Connected Wearable Motion Sensors to Assess Postoperative Mobilization. JMIR Mhealth Uhealth. 2015 Jul 28;3(3):e78. doi: 10.2196/mhealth.3785. PMID 26220691
- [Background] Cook DJ, Thompson JE, Prinsen SK, Dearani JA, Deschamps C. Functional recovery in the elderly after major surgery: assessment of mobility recovery using wireless technology. Ann Thorac Surg. 2013 Sep;96(3):1057-61. doi: 10.1016/j.athoracsur.2013.05.092. PMID 23992697
- [Background] van der Meij E, van der Ploeg HP, van den Heuvel B, Dwars BJ, Meijerink WJHJ, Bonjer HJ, Huirne JAF, Anema JR. Assessing pre- and postoperative activity levels with an accelerometer: a proof of concept study. BMC Surg. 2017 May 12;17(1):56. doi: 10.1186/s12893-017-0223-0. PMID 28494785
- [Background] Gualtieri L, Rosenbluth S, Phillips J. Can a Free Wearable Activity Tracker Change Behavior? The Impact of Trackers on Adults in a Physician-Led Wellness Group. JMIR Res Protoc. 2016 Nov 30;5(4):e237. doi: 10.2196/resprot.6534. PMID 27903490
- [Background] Paul SS, Tiedemann A, Hassett LM, Ramsay E, Kirkham C, Chagpar S, Sherrington C. Validity of the Fitbit activity tracker for measuring steps in community-dwelling older adults. BMJ Open Sport Exerc Med. 2015 Jul 8;1(1):e000013. doi: 10.1136/bmjsem-2015-000013. eCollection 2015. PMID 27900119
- [Background] Wolk S, Meissner T, Linke S, Mussle B, Wierick A, Bogner A, Sturm D, Rahbari NN, Distler M, Weitz J, Welsch T. Use of activity tracking in major visceral surgery-the Enhanced Perioperative Mobilization (EPM) trial: study protocol for a randomized controlled trial. Trials. 2017 Feb 21;18(1):77. doi: 10.1186/s13063-017-1782-1. PMID 28222805
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations for studies involving linear regression. Control Clin Trials. 1998 Dec;19(6):589-601. doi: 10.1016/s0197-2456(98)00037-3. PMID 9875838